CLINICAL TRIAL: NCT03774615
Title: A Phase IV Study to Explore the Safety of ORal IrON Supplementation With Ferric Maltol in Treating Iron Deficiency in Patients With Heart Failure Carrying Left Ventricular Assist Devices (ORION-LVAD-1)
Brief Title: ORal IrON Supplementation With Ferric Maltol in Patients With Heart Failure Carrying Left Ventricular Assist Devices
Acronym: ORION-LVAD-1
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: low recruitment rate; difficulties to achieve planned number of participants within reasonable time frame
Sponsor: Hannover Medical School (Other)
Collaborators: Shields, Shields and Associates (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORION-LVAD-1
Record Dates: First submitted 2018-12-12; First posted 2018-12-13 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2019-03

CONDITIONS: Heart Failure, Left Sided; Anemia, Iron Deficiency
Keywords: Iron Deficiency
MeSH Terms: conditions — Heart Failure; Anemia, Iron-Deficiency; Iron Deficiencies | interventions — ferric maltol

STUDY DESIGN:
Intervention Model Description: open-label, uncontrolled, monocenter, phase IV study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ferric maltol 30 mg (Feraccru®) (Experimental): Treatment with Feraccru® 30 mg hard capsules (Ferric maltol 30 mg). One capsule twice daily, morning and evening, on an empty stomach for 12 weeks
  Interventions: Drug: Ferric maltol 30 mg (Feraccru®)

INTERVENTIONS:
Drug: Ferric maltol 30 mg (Feraccru®) — Feraccru® 30 mg hard capsules will be used. Each capsule contains 30 mg iron (as ferric maltol), 91.5 mg of lactose, 0.5 mg of Allura Red AC (E129) and 0.3 mg Sunset Yellow FCF (E110) as excipients with known effects

SUMMARY:
This is a open-label, uncontrolled, monocenter, phase IV study. The aim of this study is to detect AEs or SAEs with a relative frequency of at least 11.5% in LVAD patients with iron deficiency anemia treated with oral ferric maltol for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent prior to any study-related procedure and willingness to comply with treatment and follow-up procedures
2. Male and female patients ≥18 years at day of inclusion
3. Patients capable of understanding the investigational nature, potential risks and benefits of the clinical trial
4. Patients that have an LVAD implanted for chronic heart failure and which are clinically stable for at least 6 months after LVAD implantation in the opinion of the investigator
5. 6 min walk distance >50 m
6. Mild-to-moderate iron-deficiency anemia as defined by a hemoglobin concentration ≥7 g/dl and <12 g/dl in females or ≥8 g/dl and <13 g/dl in males, and serum ferritin <100 µg/l, or 100-300 µg/l and transferrin saturation <20% at screening
7. Women of childbearing potential must:

Have a negative pregnancy test at screening Agree to use reliable methods of contraception during the course of the study

Exclusion Criteria:

1. Active hematological disorders other than iron-deficiency anemia
2. Other medical condition that according to the investigator's assessment is causing or contributing to anemia
3. Active malignancy
4. Active infectious disease
5. Active bleeding
6. Severe renal insufficiency (requiring dialysis)
7. Severe liver injury as indicated by serum aminotransferases >3 x upper limit of normal or bilirubin levels >50 µmol/l
8. Ongoing oral or intravenous iron supplementation
9. Concomitant erythropoietin medication
10. Pregnancy or lactation period
11. Subject has received any investigational medication or any investigational devices within 30 days prior to the first dose of study medication or is actively participating in any investigational drug/ devices trial, or is scheduled to receive investigational drug/devices during the course of the study.
12. Known or suspected hypersensitivity to any of the active substances or any excipients of the investigational medicinal product
13. Known haemochromatosis or other iron overload syndromes
14. Patients who have been receiving repeated (>1) blood transfusions during the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2019-11-29 (Actual)

PRIMARY OUTCOMES:
To detect AEs and SAEs with a relative frequency of at least 11.5% in LVAD patients with iron deficiency anemia treated with oral ferric maltol for 12 weeks | baseline to week 12

SECONDARY OUTCOMES:
Change in hemoglobin level from baseline to week 12 | baseline to week 12
Change in hemoglobin level from baseline to week 6 | baseline to week 6
Change in serum ferritin levels and transferrin saturation from baseline to week 6 | baseline to week 6
Change in serum ferritin levels and transferrin saturation from baseline to week 12 | baseline to week 12
Change in 6 min walking distance from baseline to week 12 | baseline to week 12
Change in serum NT-proBNP from baseline to weeks 6 | baseline to weeks 6
Change in serum NT-proBNP from baseline to weeks 12 | baseline to weeks 12
Change in echocardiographic markers of right ventricular function (right atrial area, right ventricular diameter, fractional area change, tricuspid annular plane systolic excursion) | change from baseline to week 12
Change in echocardiographic markers of left ventricular function (left ventricular ejection fraction, left atrial area, left ventricular diameter, fractional area change, tricuspid annular plane systolic excursion) | change from baseline to week 12
Liver: Change in Albumin, ALT, AST and Bilirubin from baseline to week 12 | from baseline to week 12
Liver: Change in Albumin, ALT, AST and Bilirubin from baseline to week 6 | from baseline to week 6
Kidney: Change in Creatinine (+GFR) and Urea from baseline to week 12 | from baseline to week 12
Kidney: Change in Creatinine (+GFR) and Urea from baseline to week 6 | from baseline to week 6
Change in NYHA from baseline to week 12 | from baseline to week 12

CONTACTS AND LOCATIONS:
Overall Officials: Jan Schmitto, Prof. MD, Principal Investigator — Hannover Medical School
Locations (1):
- Medizinische Hochschule Hannover, Klinik für Herz-, Thorax-, Transplantations- und Gefäßchirurgie (HTTG), Hanover, Germany